CLINICAL TRIAL: NCT00435682
Title: To Study the Peripheral Effect of Botulinum Toxin-A (Botox-A) on Experimentally Induced Cutaneous Pain in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2006-001251-35
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: The trial is performed on healthy normal males.
MeSH Terms: interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botox (Allergan Inc., US)

SUMMARY:
This is a human trial to study the peripheral effect of therapeutic botulinum toxin (botox-A). The trial is performed on healthy normal males. The study comprises of two parallel placebo-controlled, double blinded studies.

In experiment 1 intramuscular Botox will be given in corrugator (one site) and frontalis (two sites) muscles on one side and placebo to the other side. Intradermal (i.d.) capsaicin injection will be given to both sides (between the two sites of frontalis injection horizontally). Capsaicin-induced pain intensity and flare together with the area of hypersensitivity to different stimulus modalities will be measured and mapped at specific time points using different cutaneous stimuli (thermal, electrical, tactile, pressure). This will characterize which fibres and receptors are affected by Botox and will show if Botox have a unilateral effect (peripheral) or if it also affects the contralateral side (central effect).

In experiment 2 intradermal Botox will be given in corrugator (one site) and frontalis (two sites) muscles on one side and placebo to the other side. I.d. capsaicin injection will be given to both sides (between the two sites of frontalis injection horizontally). Capsaicin-induced pain intensity and flare together with the area of hypersensitivity to different stimulus modalities will be measured and mapped at specific time points using different cutaneous stimuli (thermal, electrical, tactile, pressure). This will characterize which fibres and receptors are affected by Botox. The effect of intradermal Botox will be compared to the results of experiment 1.

The two experiments will show if the intramuscular Botox exerts its action via a leak of Botox from the muscle to the overlying skin.

Antipruritic effects of Botox on histamine prick test and itch will also be assessed in parallel with the experiment 2. In this sub-experiment, 5 Units of Botox will be injected intradermally in the middle of volar forearm. The same volume of placebo will be injected into the other side. Histamine prick test will induce itch and the effect of intradermal Botox will be assessed compared to the baseline. Flare area and visual analogue scale (VAS) ratings will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Written Informed Consent
2. Male, 18 40 years of age
3. No concomitant medical diseases or clinically significant abnormal findings based on the medical history and baseline physical examination, that could affect the conduct of the study, analysis of the data, or the safety of a subject, as determined by the investigator.
4. In the opinion of the investigator, the subject clearly understands the intent of the study and is willing and able to comply with study instructions, is available for study visits and procedures and is anticipated to complete the entire study

Exclusion Criteria:

1. Any medical condition that may put the subject at increased risk with exposure to Botox, such as myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis or any other significant disease that might interfere with neuromuscular function, including peripheral neuropathies.
2. Concurrent use or use within 30 days of screening of aminoglycoside antibiotics, curare like agents or other agents that might interfere with neuromuscular function
3. Known allergy or sensitivity to any of the ingredients in the study medication or any clinical supply materials.
4. Current or previous participation in another investigational drug or device study within 30 days prior to screening.
5. Current or previous use of any serotype of botulinum toxin, or anticipated need for treatment with or use of any serotype of botulinum toxin during the study (other than the study medication).
6. Recent history of drug or alcohol abuse.
7. Indications which in the investigator's opinion, indicates inappropriate/illicit substance abuse, an underlying significant medical condition or which might interfere with the subject's participation in the study.
8. Infection or dermatological condition at the sites of study medication injection or test site.
9. Family history of hereditary neuropathy.
10. Any disease associated with a peripheral neuropathy (diabetes, etc.)
11. Anticipated need for a medical procedure, surgery or overnight hospitalization during the study
12. Concurrent use of any drug

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To determine the peripheral effect of Botox on capsaicin induced pain and related vasomotor responses.

SECONDARY OUTCOMES:
To determine which peripheral nociceptors (pain sensitive nerve endings) are blocked by Botox.
To determine the effect of intradermal Botox on itch.

CONTACTS AND LOCATIONS:
Overall Officials: Lars - Arendt-Nielsen, Prof., Dr.Med.Sci., Ph.D., Study Chair — Aalborg University, Center for Sensory-Motor Interaction (SMI); Asbjoern Mohr Drewes, MD, PhD, DMSc, Prof., Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

REFERENCES:
- [Background] Gazerani P, Staahl C, Drewes AM, Arendt-Nielsen L. The effects of Botulinum Toxin type A on capsaicin-evoked pain, flare, and secondary hyperalgesia in an experimental human model of trigeminal sensitization. Pain. 2006 Jun;122(3):315-325. doi: 10.1016/j.pain.2006.04.014. Epub 2006 May 4. PMID 16677761